CLINICAL TRIAL: NCT05118867
Title: Improve the Patients' Recovery by Engagement and Partnerships With Family- CaregiveRs to End Delirium (iPREPARED) - A Feasibility and Acceptability Study
Brief Title: Improve the Patients' Recovery With Family- Caregivers to End Delirium
Acronym: iPREPARED
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: To update technology based on feedback from participants
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Heidi L. Lindroth PhD RN, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-005022
Record Dates: First submitted 2021-10-08; First posted 2021-11-12 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Delirium
Keywords: Aged 60 years old or older; Hospitalized with a risk of confusion; At risk of falling; At risk of vision or hearing impaired
MeSH Terms: conditions — Delirium; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPREPARED Hospital Recovery Club (Experimental): Participants and their recovery partners (informal caregivers) will use the iPREPARED mobile health technology. They will watch a short video to prepare them for their hospital stay and asked to use the provided resources and tools to maintain their brain health during their hospital stay.
  Interventions: Behavioral: iPREPARED
- Standard Hospital Care Group (No Intervention): Participants will receive standard protocolized care procedures.

INTERVENTIONS:
Behavioral: iPREPARED — iPREPARED is a mobile health technology that can be accessed via the web, tablet, or phone. It contains a preparatory video that outlines what to expect during the hospitalization. Instructional videos and examples are provided for the patient and their recovery partner to use to do their own reorientation, distraction techniques, physical activity, and sleep hygiene.
  Arms: IPREPARED Hospital Recovery Club

SUMMARY:
This research is being done to find out if patients and caregivers who use the iPREPARED mobile health technology experience less delirium, a type of acute confusion, and if they do experience delirium, the delirium will be less severe and distressful.

iPREPARED prepares patients and caregivers on what to expect during their hospital stay and provides instructions and resources on how to use non-pharmacologic strategies like re-orientation, distraction techniques, and other activities to maintain their brain health during their hospital stay.

DETAILED DESCRIPTION:
The purpose of this pilot study is to assess the feasibility, acceptability, and preliminary efficacy of the iPREPARED mobile health technology to reduce delirium incidence in a two-group, pilot randomized- controlled clinical trial. In the context of this intervention, the caregiver is defined as a patient-identified family member or friend that can accompany the patient in their hospital journey.

Aim 1: Determine the feasibility, acceptability, and usability of the iPREPARED intervention for use by older hospitalized adults (>60yo) and their caregivers (patient-caregiver dyad).

Aim 2: To estimate the effect size needed to reduce the incidence of delirium in participants using the iPREPARED intervention.

Aim 3: Identify patient-caregiver reported strategies to improve the usability of the iPREPARED intervention.

Secondary Outcomes:

1. Association between delirium incidence and self-rated health status (GSRH).
2. Association between delirium incidence, severity, and delirium-related distress (NCCN Distress thermometer) and resiliency (BRS resiliency scale).
3. Acute stress measured by the IPAT will be compared across the two groups. Acute stress measured by the Intensive Care Psychological Assessment Tool (IPAT) will be less in the intervention group.
4. Delirium-related distress will be analyzed across the two groups. Delirium-related distress measured by the NCCN Distress Thermometer will be less in the intervention group.
5. Plasma and serum biomarker differences between groups and between delirium/non- delirium cohort.
6. Clinical outcomes including adverse hospital events (falls, nosocomial infections, aspirations), length of hospital stay, discharge disposition, mortality and 30-day readmission rates will be collected and examined between groups:

   1. Nosocomial infection is defined as a diagnosis not present on admission and occurred after 48 hours of hospital admission and includes UTI, Pneumonia, Decub ulcers, Cellulitis, CAUTI's and CLABSI's

ELIGIBILITY:
Patient Inclusion Criteria:

* 60 years of age or older
* Have 1 risk factor for delirium (pre-existing cognitive impairment, vision/hearing impairment, identified as high risk for falls, illness rated as severe)
* Estimated length of stay of 24 hours or more in hospital
* Have an informal caregiver (18 years of age or older, family member or friend) willing to participate

Patient Exclusion Criteria:

* Patient lacks capacity to consent
* Unable to communicate or participate in study due to language barriers or sensory deficits
* Prisoners
* Documented history of dementia in the medical record
* Patient admitted to hospice service or actively dying
* Delirium present upon admission to hospital
* COVID-19 positive test

Caregiver Inclusion Criteria:

* 18 years of age or older
* Family member, friend, or neighbor of the patient willing to participate in the study and support the patient during the study period (support can be in-person or virtual)

Caregiver Exclusion Criteria:

- Unable or unwilling to participate due to language barriers, availability, or other communication barriers

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study recruitment to intervention study | Number approached for study that were eligible and number consented into study over 2-year study.
  Total number of patient-caregiver dyads enrolled in the study
Usability and acceptability of digital technology | From enrollment through study completion, an average of 4 days
  Measured using the System Usability Scale and the treatment acceptability preference questionnaire which measure the participants self-reported usability and acceptability of the iPREPARED intervention.
Delirium incidence | From enrollment through study completion, an average of 4 days
  The incidence of delirium will be assessed upon enrollment then twice daily on days 1-4 of the study, and upon hospital discharge using the 3DCAM. Effect sizes between groups will be generated for future larger studies.

SECONDARY OUTCOMES:
Delirium-related distress | From enrollment through study completion, an average of 4 days
  The NCCN distress thermometer will be used twice daily to assess the level of self-reported distress associated with the signs and symptoms of delirium.
Resiliency | At enrollment into study
  Measured using the brief resilience scale that assesses the participants ability to recover from stressful events through 6-item questionnaire asking participants to response to questions on a scale of strongly disagree, disagree, neutral, agree, or strongly agree.
General Self-Rated Health Status | At enrollment into study
  Measured using the self-reported general self-rated health status (GSRH) asking participants to rate their general health as good, rather good, poor, or very poor.
Delirium Severity | From enrollment through study completion, an average of 4 days
  Delirium severity will be assessed using the Delirium Rating Scale - R- 98 (DRS-R-98). This will be assessed upon enrollment, twice daily on hospital days 1-4, and upon discharge.
Acute Stress associated with the hospitalization | From enrollment through study completion, an average of 4 days
  The Intensive Care Psychological Assessment Tool (IPAT) will be administered with concurrent delirium incidence and severity measurement.47 This is a 10-item scale that evaluates how a patient has been feeling since their admission. These answers will inform the delirium assessments.
Biomarkers | At enrollment and Day 4
  Plasma and serum biomarker differences between groups and between delirium/non-delirium cohort
Discharge disposition | From enrollment through study completion, an average of 4 days
  Place (home, rehabilitation facility, long term care facility) that patient was discharged from the hospital to for continued care.
30-day readmission rates | 30-days after hospital discharge date
  Rate of patients that were re-admitted to the hospital following the index hospitalization
Length of hospital stay | From enrollment through study completion, an average of 4 days
  Number of days admitted to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Lindroth, PhD, RN, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with the NIDUS network and for other interested investigators. Please contact study team.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: November 1 2021-December 31 2023
Access Criteria: Email investigator